CLINICAL TRIAL: NCT01951391
Title: Effect of Surfactants on the Skin Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tissa Hata, MD, MD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCSD 111296
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Healthy Skin
Keywords: study; subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Soap vs. Benzalkonium Chloride Soap (Other): Each subject's will have one forearm washed with a control soap and then the other forearm will be washed with benzalkonium chloride soap. The control forearm will be swabbed for bacteria at baseline, 10 minutes, 6 hours, and 24 hours. The benzalkonium chloride forearm will be swabbed at baseline and 6 hours.
  Interventions: Other: Control Hand Soap; Other: Benzalkonium Chloride Soap
- Control Soap vs. Triclocarban Soap (Other): Each subject's will have one forearm washed with a control soap and then the other forearm will be washed with triclocarban soap. The control forearm will be swabbed for bacteria at baseline, 10 minutes, 6 hours, and 24 hours. The triclocarban forearm will be swabbed at baseline and 6 hours.
  Interventions: Other: Control Hand Soap; Other: Triclocarban Soap

INTERVENTIONS:
Other: Control Hand Soap — Commercially available soap will be used to wash the subject's forearms
Other: Benzalkonium Chloride Soap — Commercially available soap containing benzalkonium chloride will be used to wash the subject's forearms
  Arms: Control Soap vs. Benzalkonium Chloride Soap
Other: Triclocarban Soap — Commercially available soap containing triclocarban will be used to wash the subject's forearms
  Arms: Control Soap vs. Triclocarban Soap

SUMMARY:
Up to 10 volunteers will be recruited to evaluate the microbial environment on their forearms. Following informed consent, bacterial swabs will be obtained at baseline from the forearms of all subjects. Their forearms will then be washed with one of the study cleansers. Subjects will then have their forearms swabbed for bacteria at the following time points: 10 minutes, 6 hours, and 24 hours after the wash. DNA will be extracted from all swabs and bacterial diversity evaluated by 16S pyrosequencing.

DETAILED DESCRIPTION:
The timeline for the patients will be as follows:

On Day 0, after being given a witnessed, written, informed consent, a medical history and a limited physical exam will be performed. If using certain topical products and medications that are not allowed during this study, patients may be asked to withhold them for the remainder of the study. The study doctor or study coordinator will explain which medications and activities are not allowed during this study. Baseline bacterial swabs from the bilateral volar forearms will be collected followed by application and rinsing of a hand wash with an antimicrobial compound (benzalkonium chloride or triclocarban) on the right forearm, and a cleanser without an antimicrobial compound (control) on the left forearm. 200 microliters of water/hand wash will be applied to the volar forearms and lather generated for 15 seconds using a gloved hand. The lather will be allowed to stay in contact with the skin for an additional 30 seconds. The total contact time will be 60 sec. The forearm will be rinsed with running tap water for 15 seconds, air-dried for 5 minutes and the skin surface will again be swabbed for bacteria 10 minutes after the wash. The same procedure will be repeated on the 2nd volar forearm with the opposing wash. Subjects will then have repeat skin swabs at 6 hours +/- 1 hour and at 24 hours +/- 6 hours after washing. Subjects will be instructed to avoid rigorous exercise/swimming, significant sun exposure (i.e. sunbathing), cleaning the forearms with other antibacterial products, and showering during these 24 hours.

ELIGIBILITY:
Inclusion Criteria:

Those who meet all of the following criteria are eligible for enrollment into the study:

1. Age 18-60 years
2. Male or female of any race and ethnicity
3. Subject agrees to comply with study requirements.

Exclusion Criteria:

1. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
2. Dermatologic disease such as psoriasis or atopic dermatitis which may have inherently abnormal antimicrobial peptide levels
3. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
4. Pregnant or nursing females
5. Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
6. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
7. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
8. Active viral or fungal skin infections at the target areas
9. Are currently receiving lithium, antimalarials, or intramuscular gold now or within the last 4 weeks.
10. Ongoing participation in an investigational drug trial
11. Use of any oral or topical antibiotic during the study and up to one week prior to entering the study
12. Use of any local topical medications less than one week prior to screening
13. Use of any systemic immunosuppressive therapy less than four weeks prior to screening.
14. Subjects with a history of or propensity to developing reactions after use of over the counter cleansers
15. Subjects with diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Soap vs. Benzalkonium Chloride Soap | Control Soap vs. Triclocarban Soap
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Forearms
Groups:
- Control Soap vs Benzalkonium Chloride Soap: Each subject's will have one forearm washed with a control soap and then the other forearm will be washed with benzalkonium chloride soap. The control forearm will be swabbed for bacteria at baseline, 10 minutes, 6 hours, and 24 hours. The benzalkonium chloride forearm will be swabbed at baseline and 6 hours.
- Control Soap vs Triclocarban Soap: Each subject's will have one forearm washed with a control soap and then the other forearm will be washed with triclocarban soap. The control forearm will be swabbed for bacteria at baseline, 10 minutes, 6 hours, and 24 hours. The triclocarban forearm will be swabbed at baseline and 6 hours.
- Total: Total of all reporting groups
Arm/Group | Control Soap vs Benzalkonium Chloride Soap | Control Soap vs Triclocarban Soap | Total
Number analyzed (Participants) | 5 | 5 | 10
Number analyzed (Forearms) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 34 [29 to 36] | 31.8 [25 to 38] | 32.9 [25 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative 16S Abundance - Control Soap
Description: Total bacterial DNA abundance at baseline (relative to baseline), prior to washing with control soap (softsoap aquarium series hand soap) as measured by qPCR of 16S RNA
Time Frame: Baseline, 10 minutes, 6 hours, 24 hours
Population: The control soap data for all 10 subjects (5 from each treatment arm) was pooled for this analysis. The control soap subjects' forearms were were assessed at the following time points--baseline, 10 minutes, 6 hours, and 24 hours.
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Groups:
- Control Hand Soap: Prior to washing, each subjects' forearms will be swabbed for bacteria. Each subject will then be washed with Softsoap aquarium series hand soap. They will then be swabbed at 10 minutes, 6 hours, and 24 hours to determine changes in bacteria levels.
Arm/Group | Control Hand Soap
Number analyzed (Participants) | 10
Percentage of Baseline
  Baseline | 100 [100 to 100]
  10 Minutes | 74 [58 to 110]
  6 Hours | 84 [58 to 680]
  24 Hours | 100 [42 to 680]

2. Secondary Outcome: Relative Abundance of Staphylococcus Epidermidis of Intervention Arms
Description: Total bacterial DNA abundance of S. epidermidis (relative to baseline) at baseline and 6 hours, before washing with any soap as measured by qPCR of 16S RNA
Time Frame: Baseline, 6 hours
Population: The control soap data for all 10 subjects (5 from each treatment arm) was pooled for this analysis. The control soap subjects' forearms were were assessed at the following time points--baseline and 6 hours. The benzalkonium chloride and triclocarban forearms were assessed at the same time points.
Measure: Mean (Standard Error); unit: Percentage of Baseline
Groups:
- Control Hand Soap: Prior to washing, each subjects' control soap forearm will be swabbed for bacteria. Each subject will then be washed with Softsoap aquarium series hand soap. They will then be swabbed at 6 hours to determine changes in staphylococcus epidermidis levels.
- Benzalkonium Chloride Soap: Prior to washing, each subject's benzalkonium chloride forearm will be swabbed for bacteria. Each subject will then be washed with a soap containing benzalkonium chloride. They will then be swabbed at 6 hours to determine changes in staphylococcus epidermidis levels.
- Triclocarban Soap: Prior to washing, each subject's triclocarban forearm will be swabbed for bacteria. Each subject will then be washed with a soap containing triclocarban. They will then be swabbed at 6 hours to determine changes in staphylococcus epidermidis levels.
Arm/Group | Control Hand Soap | Benzalkonium Chloride Soap | Triclocarban Soap
Number analyzed (Participants) | 10 | 5 | 5
Percentage of Baseline
  Baseline | 100 (0) | 100 (0) | 100 (0)
  6 Hours | 283 (190) | 100 (32) | 200 (150)

ADVERSE EVENTS:
Arm/Group | Control Soap vs. Benzalkonium Chloride Soap | Control Soap vs. Triclocarban Soap
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No